CLINICAL TRIAL: NCT06640556
Title: The Effect of "Green Future With Midwife Hands" Climate Change Animation on Mothers' Climate Change Awareness and Behavior
Brief Title: The Effect of"Green Future With Midwife Hands"Climate Change Animation on Mothers' Climate Change Awareness and Behavior
Acronym: RKÇ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Senem Çiçek, Master of Degree, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-SBT-SÇ-1
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Climate Change; Awareness; Conscious; Consumption; Consumption Habits of Mothers
Keywords: Climate change; awareness; conscious; consumption; consumption habits of mothers

STUDY DESIGN:
Intervention Model Description: The group that watched the animation and the group that did not watch it
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will be blinded in the study. The researcher will not be blinded because he/she is the implementer. However, the researcher will open the envelope created by the statistician just before the application and learn which group the mother is in. In order to prevent bias in the evaluation of the data, the groups will be coded as A and B, and the data will be analysed by an independent statistician. After the analysis and interpretation of the data is completed, the codes of the intervention and control groups will be revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-intervention group (No Intervention): the group will not be trained
- Mothers who have had a caesarean section or normal birth (Experimental): The animation "A Green Future with the Hands of a Midwife" will be downloaded to mothers' phones and played in a quiet and non-stimulating environment before discharge. In addition, the animation will be played again after the data collection tools are applied on the 7th, 21st and 30th day.
  Interventions: Behavioral: watching animation show

INTERVENTIONS:
Behavioral: watching animation show — The intervention group will watch the animation titled 'A Green Future with the Hand of a Midwife' on days 7, 21, and 30 to mothers who have just given birth, and the scale will be evaluated on three separate days in total.
  Other Names: pre-test data (animation show) ,post- test 7. day,21 and 30. day
  Arms: Mothers who have had a caesarean section or normal birth

SUMMARY:
The Effect of "Green Future with Midwife Hands" Climate Change Animation on Mothers' Climate Change Awareness and Behavior Climate change appears as one of the most important environmental problems of today. Many negative effects such as the increase in greenhouse gas emissions, global warming, sea level rise and the frequency of extreme weather events threaten both natural ecosystems and human life. In this context, it is of great importance for individuals to gain awareness about climate change and exhibit environmentally friendly behavior for a sustainable future. In particular, mothers and expectant mothers have the potential to create significant awareness and change by choosing products that do not harm the environment, while looking for the best for their babies. Reducing plastic use, choosing organic textile products, using biodegradable wet wipes and choosing toys made from natural materials both protect babies' health and support environmental sustainability. This awareness reinforces the environmentally friendly behavior of mothers and helps future generations grow up as more conscious individuals. The role of mothers in this regard is undeniably great for a sustainable future. While mothers making environmentally friendly choices increases the environmental awareness of not only their own families but also the wider masses, being careful when choosing carbon footprint baby products both protects the health of babies and reduces environmental impacts.

This research aims to encourage mothers and expectant mothers to make environmentally friendly and carbon footprint-reducing choices when choosing baby products by increasing the climate change awareness of mothers and expectant mothers through the "Green Future with Midwife Hands" Climate Change Animation.

DETAILED DESCRIPTION:
Climate change is one of the most important ecological problems of the 21st century, which causes global warming due to the accumulation of greenhouse gases in the atmosphere resulting from human activities. This situation creates serious effects on economic, social, environmental and health. Women, especially in developing countries, are more affected by climate change; when water and food security decreases, these responsibilities make them more vulnerable socially and economically. This project aims to raise awareness of climate change for mothers through animation-based education and to encourage them to prefer nature-friendly baby products. It also aims to contribute to leaving a cleaner future for nature by providing guidance to mothers on the correct management of waste. The project has unique value as it is the first animation education model specialized for mothers in Turkey and contributes to sustainable development goals.

ELIGIBILITY:
Inclu• Pregnant women who can read and write Turkish,

* Volunteer to participate in the research,
* Have had a normal or cesarean delivery,
* Are primiparous,
* Are open to communication (able to understand and answer questions) will be included in the samplesion Criteria:

Exclusion Criteria:

* • Those who do not have the ability to read, listen, write, speak and understand Turkish,

  * Those who have hearing or visual impairments,
  * Those who have postpartum complications,
  * Those who have had a stillbirth,
  * Those who wish to withdraw from the study were not included.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who have given birth normally or by cesarean section, Primiparous,Those who are open to communication (able to understand and answer questions)
Enrollment: 666 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Scale for Assessing Mothers' Behaviors Towards Climate Change | 7,21 and 30. day
  In order to determine the behaviors of mothers towards climate change, a scale will be prepared to evaluate the use of washable diapers, environmentally friendly diapers and disposal of waste diapers, selection of baby textile products and excess textile consumption and disposal, use and disposal of baby bottles, pacifiers and plastic products, selection of wooden toys instead of plastic toys, and the effects of microplastics on baby health.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Ünivesitesi tıp fakültesi hastanesi, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
YES
Supporting Information: Study Protocol
Time Frame: 10/09/2025 - 15/06/2025